CLINICAL TRIAL: NCT00240292
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group, Multicentre, Phase III Study to Assess the Impact of Rosuvastatin Treatment for 26 Weeks (Titrated to a Maximum Dose of 40mg Once Daily) on Left Ventricular Function, Cytokines and Lipid Parameters in Patients With Established Systolic Chronic Heart Failure.
Brief Title: Rosuvastatin Impact on Ventricular Remodelling Lipids and Cytokines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4522AS/0002
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Heart Failure, Congestive
Keywords: Ischaemic or non-ischaemic systolic congestive heart failure
MeSH Terms: conditions — Heart Failure; Ischemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor

SUMMARY:
The purpose of this study is to assess the effect of rosuvastatin (up-titrated to a dose of 40mg/day) compared to placebo on cardiac remodelling, estimated by change in left ventricular ejection fraction on radionuclide ventriculography, at 26 weeks post randomisation from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, males or females aged 18 or older, LVEF ≤ 40% assessed by RNVG or contrast ventriculogram or ≤ 35% assessed by TTE within the previous 6 months, LVEF < 45% as assessed by RNVG during Visit 1, NYHA Class II, III or IV symptoms primarily related to heart failure, ischaemic and non-ischaemic patients and on stable heart failure therapy as defined by physician's best practice.

Exclusion Criteria:

* Key exclusion criteria include acute myocarditis within the last 12 months, diabetes mellitus not controlled by diet, oral therapy or insulin therapy, homozygous familial hypercholesterolaemia, receiving biventricular pacing or expected to receive biventricular pacing in the next 6 months, subjects who normally would be considered for statin therapy in the next 6 months, sever hypertension, history of definite myocardial infarction, cerebrovascular accident, percutaneous transluminal coronary angioplasty or coronary bypass graft within 3 months prior to enrolment in the study, body mass index < 15, plus others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2003-02

PRIMARY OUTCOMES:
Determine the effect of rosuvastatin (up-titrated to a dose of 40mg/day) compared to placebo on cardiac remodelling, estimated by change in left ventricular ejection fraction on radionuclide ventriculography, at 26 weeks post randomization from baseline.

SECONDARY OUTCOMES:
Determine the effects of rosuvastatin (up-titrated to a dose of 40mg/day) compared to placebo by measuring:
Changes from baseline at 26 weeks post-randomisation, of left ventricular (LV) end-diastolic and end-systolic diameter, and LV fraction shortening, as determined by transthoracic echocardiography.
The percentage change in lipid parameters: total cholesterol, low density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides after 6, 12 and 26 weeks post-randomisation
Changes from baseline at 26 weeks post-randomisation in neurohormonal and immunological markers: norepinephrine, endothelin, N-terminal pro-brain natriuretic peptide, high-sensitivity C-reactive protein, tumour necrosis factor α and interleukin 6.
Assess the safety of rosuvastatin over 26 weeks determined by the incidence and severity of adverse events and abnormal laboratory values.
Assess change in quality of life score, as determined by the Minnesota Living with Heart Failure questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS PhD FRACP, Principal Investigator — Clinical Pharmacology, Department of Epidemiology and Preventative Medicine, Monash University, Alfred Hospital
Locations (13):
- Australia (13):
  - Research Site, Canberra, Australian Capital Territory
  - Research Site, Gosford, New South Wales
  - Research Site, Newcastle, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Nambour, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Launceston, Tasmania
  - Research Site, Geelong, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Mildura, Victoria
  - Research Site, Perth, Western Australia